CLINICAL TRIAL: NCT06739681
Title: The Effect of Imagery and Breathing Exercises on Postural Sway and Target Achievement in Olympic Archers
Brief Title: The Effect of Imagery Exercises on Attention and Performance in Olympic Archers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Cansu Keskin, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMU-FTR-CK-01
Record Dates: First submitted 2024-06-07; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Performance Improvement in Beginner Archers
Keywords: Breathing Exercises; Imagination; Cognition; Exercise; Sports; Young Adult
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (CG) (No Intervention): Only routine exercise program will be applied
- Imagination Group (IG) (Active Comparator): In addition to routine exercises, a 15-minute visualization session will be applied.
  Interventions: Other: Routine Intervention; Other: Mental Imagery Intervention
- Respiratory Group (RG) (Active Comparator): Breathing exercises will be applied in addition to routine exercises.
  Interventions: Other: Routine Intervention; Other: Breathing Exercise Intervention

INTERVENTIONS:
Other: Routine Intervention — These routine exercises used in archery training will be applied to all participants. Exercise sessions will be planned 2 days a week, every other day, for 8 weeks. It will progress progressively according to the athlete's tolerance.
  Arms: Imagination Group (IG); Respiratory Group (RG)
Other: Mental Imagery Intervention — Mental Imagination will be done with Recording Audio. An audio recording will last 5 minutes. The audio recording will be listened to 3 times in one session. The total visualization session will last 15 minutes in a dark and quiet room.
  Arms: Imagination Group (IG)
Other: Breathing Exercise Intervention — Participants participating in Pranayama training will practice in a comfortable position in a quiet room at a temperature of 25 ± 2°C. The slow pranayama technique chosen is alternate nasal breathing (Nadishodhana Pranayama).
  Arms: Respiratory Group (RG)

SUMMARY:
The goal of this clinical trial is to for beginners in archery in to examine the effects of Imagination and breathing exercises given in addition to 8-week archery training on archery target score, postural sway, attention, hand grip, visualization and respiratory function parameters.. The main questions it aims to answer are:

* Do Imagination and breathing exercises have an effect on archery target shooting score?
* Do breathing exercises positively affect shooting performance by reducing postural sway?
* Do archers' imagination skills positively affect their attention and performance?
* Do hand grip strength and reaction time positively affect shooting performance?

Participants will Routine exercises used in archery training will be applied to all participants.

Researchers will compare control group, Imagination group and meditation group to see if Control group (CG); Only routine exercise program will be applied. To the Imagination Group (IG); In addition to routine exercises, a 15-minute visualization session will be applied. Respiratory Group (SG); Breathing exercises will be applied in addition to routine exercises.

ELIGIBILITY:
Inclusion Criteria:

* Completing the study consent form,
* Successful in the The Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST),
* Successful in the Upper Quarter Y Balance Test (YBT),
* Those who do archery sports were included in the study.

Exclusion Criteria:

* Having musculoskeletal system problems,
* Having a neurological disease,
* Having vestibular disease,
* Having pulmonary disease,
* Hearing loss,
* Those who have undergone orthopedic surgery will not be included in the study.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Postural Sway Assessment | Day 1 and 8 weeks later
  Postural Sway Assessment will be evaluated with SWAY Medical Balance Application
Evaluation of Respiratory Function Test Parameters | Day 1 and 8 weeks later
  Evaluation of Respiratory Function Test Parameters will be done with spirometry test. FEV1, FVC, FEV1/FVC Physiological values will be recorded.
Evaluation of Archery Shooting Performance | Day 1 and 8 weeks later
  Evaluation of Archery Shooting Performance, Archery Shooting Performance Test will be used to measure shooting performance.

SECONDARY OUTCOMES:
Hand Grip Strength | Day 1 and 8 weeks later
  Hand Grip will be measured with Jamar hand dynamometer
Reaction Time | Day 1 and 8 weeks later
  Reaction Time will be done from Human Benchmark website
Mental Imagery Assessment | Day 1 and 8 weeks later
  Mental Imagery Assessment will be done with the Mental Training Inventory in Sports

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The protocol of the exercises will be shared according to the weeks.
Supporting Information: Study Protocol
Time Frame: 6 months after publication.

REFERENCES:
- [Background] Spratford W, Campbell R. Postural stability, clicker reaction time and bow draw force predict performance in elite recurve archery. Eur J Sport Sci. 2017 Jun;17(5):539-545. doi: 10.1080/17461391.2017.1285963. Epub 2017 Feb 14. PMID 28276913
- [Background] Savvides A, Giannaki CD, Vlahoyiannis A, Stavrinou PS, Aphamis G. Effects of Dehydration on Archery Performance, Subjective Feelings and Heart Rate during a Competition Simulation. J Funct Morphol Kinesiol. 2020 Aug 27;5(3):67. doi: 10.3390/jfmk5030067. PMID 33467282
- [Background] Kolayiş İE, Mimaroğlu E. Okçuluk Milli Takımının Antrenman Ortamında Kalp Atım Hızı ve Nişan Alma Süresinin Atış Puanı Üzerindeki Etkileri. Uluslararası İnsan Bilimleri Dergisi. 2008;(May 2008).
- [Background] Grassmann M, Vlemincx E, von Leupoldt A, Mittelstadt JM, Van den Bergh O. Respiratory Changes in Response to Cognitive Load: A Systematic Review. Neural Plast. 2016;2016:8146809. doi: 10.1155/2016/8146809. Epub 2016 Jun 14. PMID 27403347
- [Background] Dulan J. Archery Stance And Breath Control Article in. Int J Innov Res Sci Eng Technol [Internet]. 2022; Available From: www.ijmrset.com
- [Background] Andrade DC, Melipillan C, Toledo C, Rios-Gallardo A, Marcus NJ, Ortiz FC, Martinez G, Munoz Venturelli P, Del Rio R. Heart rate and cardiac autonomic responses to concomitant deep breathing, hand grip exercise, and circulatory occlusion in healthy young adult men and women. Biol Res. 2021 Sep 26;54(1):32. doi: 10.1186/s40659-021-00355-1. PMID 34565477
- [Background] Palmer TB, Maurya PS, Sisneros KP, Palmer BM. Can handgrip strength measurements predict postural balance performance in older women? J Musculoskelet Neuronal Interact. 2023 Mar 1;23(1):36-42. PMID 36856098
- [Background] Lu Q, Li P, Wu Q, Liu X, Wu Y. Efficiency and Enhancement in Attention Networks of Elite Shooting and Archery Athletes. Front Psychol. 2021 Mar 9;12:638822. doi: 10.3389/fpsyg.2021.638822. eCollection 2021. PMID 33767650
- [Background] Yachsie BTPWB, Suharjana, Graha AS, Prasetyo Y, Nasrulloh A, Suhasto S. Mental Training to Improve the 40-Meter-Distance Archery Accuracy With Imagery and Meditation Methods. International Journal of Human Movement and Sports Sciences. 2023 Apr 1;11(2):450-6.
- [Background] Robin N, Dominique L. Mental İmagery And Tennis: A Review, Applied Recommendations and New Research Directions. Movement & Sport Sciences - Science & Motricité. 2022;
- [Background] Sharma VK, Trakroo M, Subramaniam V, Rajajeyakumar M, Bhavanani AB, Sahai A. Effect of fast and slow pranayama on perceived stress and cardiovascular parameters in young health-care students. Int J Yoga. 2013 Jul;6(2):104-10. doi: 10.4103/0973-6131.113400. PMID 23930028
- [Background] Teixeira AL, De Oliveira AS, Rodrigues NA, Bueno GAS, Novais MEO, De Paula Moreira R, et al. Reference Values, İntrarater Reliability, And Measurement Error For The Closed Kinetic Chain Upper Extremity Stability Test And Upper Quarter Y Balance Test İn Young Adults. Motriz Revista De Educacao Fisica. 2022;28.
- [Background] Mummareddy N, Brett BL, Yengo-Kahn AM, Solomon GS, Zuckerman SL. Sway Balance Mobile Application: Reliability, Acclimation, and Baseline Administration. Clin J Sport Med. 2020 Sep;30(5):451-457. doi: 10.1097/JSM.0000000000000626. PMID 29952841
- [Background] Yarayan YE, Levent E, Gazi İ. Sporda Zihinsel Antrenman Envanteri'nin (SZAE) Uyarlama Çalışması. Vol. 23, Gazi Beden Eğitimi ve Spor Bilimleri Dergisi Gazi Journal of Physical Education and Sport Sciences. 2018.
- [Background] Ersin A, Tezeren Hc, Pekyavas No, Asal B, Atabey A, Diri A, et al. The Relatıonshıp Between Reactıon Tıme and Gamıng Tıme in E-Sports Players. Kinesiology. 2022;54(1).